CLINICAL TRIAL: NCT06360068
Title: A Prospective, Single Arm, Open Label, Proof of Concept Clinical Study of Sulfasalazine in the Treatment of Active Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qiong Fu (Other)
Responsible Party: Sponsor-Investigator, Qiong Fu, Clinical professor, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLE-SASP POC; 82371767 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Sulfasalazine; interferon
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulfasalazine group (Experimental)
  Interventions: Drug: Sulfasalazine Tablets

INTERVENTIONS:
Drug: Sulfasalazine Tablets — All subjects who meet the inclusion/exclusion criteria will be given sulfasalazine 750mg/dose, twice a day. The dosage will be increased to 1000mg/dose within one month, twice a day if the patient tolerates well.

SUMMARY:
The goal of this clinical trial is to learn if sulfasalazine is safe and feasible in the treatment of active lupus erythematosus (SLE). The main questions it aims to answer are:

Does drug sulfasalazine with stable background treatment help lower the disease activity (SLEDAI) at week 16? How many patients can reach SRI-4 at week 16? Can this regimen help lower the prednisone dosage the patients need at week 16? What about the change of the type I interferon related genes expression at week 16?

Participants will:

Take sulfasalazine 750mg/dose, twice a day for 16 weeks. The dosage will be increased to 1000mg/dose within one month, twice a day if the patient could tolerate.

Visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE according to the 2012 SLICC SLE classification criteria.
* 18 to 65 years old, regardless of gender.
* Active SLE, i.e. SLEDAI-2K score ≥ 4 points at enrollment.
* Receiving standard of care:

  1. Prednisone dosage≤20mg/day, with or without hydroxychloroquine (HCQ,≤400mg/day), classic immunosuppressive agents (IS),ie, mycophenolate mofetil(≤2.0g/day), azathioprine (≤2mg/kg/day), cyclosporine(≤5.0mg/kg/day), tacrolimus(≤3.0mg/day), methotrexate(≤20mg/week), leflunomide(≤40mg/day), or biological agents such as belimumab(≤ 10mg/kg/month) and telitacicept (≤160mg/week);
  2. No more than three types of combined classic IS or biological agents, not including HCQ.
  3. Prednisone dosage should NOT be increased within one month of the screening period, and the immunosuppressants regimen should be stable for at least one month.
* Agree to sign the informed consent form.
* Agree to receive contraception through intrauterine devices or oral contraceptives (progesterone or compound progesterone) or condoms.

Exclusion Criteria:

* Severely active SLE: SLEDAI-2K >12 at screening.
* 24-hour urine protein≥ 3g/24 hours.
* eGFR < 60mL/min/1.73m2 (EPI formula).
* Baseline prednisone dosage>40mg/d at screening.
* Other autoimmune diseases, such as rheumatoid arthritis, Sjogren's syndrome, myositis, scleroderma, autoimmune liver disease, etc.
* Leukopenia or thrombocytopenia (WBC≤3×109/L or PLT≤50×109/L) not caused by SLE.
* Liver dysfunction (ALT or AST more than twice the normal upper limit).
* Allergic to sulfonamide drugs.
* Pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
the change of disease activity (SLEDAI score) | 16 weeks
  reaching the SLEDAI score based on clinical symptoms and laboratory tests according to the SLEDAI score system

SECONDARY OUTCOMES:
the number of patients who can reach SRI-4 | 16 weeks
  SRI-4 is defined as: 1.the SELENA-SLEDAI score decreased by ≥ 4 points compared to baseline, and there were no new BILAG grade A or ≤ 2 new BILAG grade B compared to baseline, and the overall physician assessment (PGA) did not deteriorate (an increase of<0.30 points from baseline)
the change of prednisone dosage | 16 weeks
  baseline prednisone dosage subtracts the prednisone dosage at week 16.

OTHER OUTCOMES:
the change of interferon stimulating genes (ISG) expression | 16 weeks
  the ISG level at baseline subtracts the ISG level at week 4, week 8, week 12 and week 16.

IPD SHARING:
Plan to Share IPD: No